CLINICAL TRIAL: NCT01066572
Title: Paramedic Initiated Lisinopril For Acute Stroke Treatment: a Pilot Randomised Controlled Trial
Brief Title: Paramedic Initiated Lisinopril For Acute Stroke Treatment
Acronym: PIL-FAST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: North East Ambulance Service NHS Foundation Trust (Other); Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP-PG-0606-1241
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Lisinopril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisinopril (Experimental): Experimental
  Interventions: Drug: Lisinopril
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisinopril — 5-10 mg Lisinopril per day for seven days, depending on blood pressure.
  Other Names: ACE inhibitor
  Arms: Lisinopril
Drug: Placebo — Matched placebo; identical tablets to Lisinopril.
  Other Names: Dummy drug
  Arms: Placebo

SUMMARY:
This study aims to investigate the use of lisinopril to lower blood pressure in stroke patients, pre-hospital, by research-trained paramedics.

DETAILED DESCRIPTION:
High blood pressure immediately following stroke is common and related to poorer stroke functional outcome and death. Although treatment of high blood pressure is well established for thre prevention of stroke, it is unclear if high blood pressure observed immediately after stroke should be lowered.

Several previous clinical trials have lowered blood pressure in acute stroke but this has not resulted in improved stroke outcome. One reason for this may be because treatment was started too late after stroke occurred. There is rapid progression of brain injury following stroke and any stroke treatment may need to be started very early to have a beneficial effect. Previous trials started blood pressure lowering after patients arrived at hospital and this was usually a significant time after stroke occurred.

The earliest time after stroke that blood pressure treatment could be started is during contact with the emergency medical services (paramedics). This research study is a pilot double blind randomised controlled trial of paramedic initiated blood pressure treatment for patients with high blood pressure immediately after stroke.

Patients with high blood pressure and suspected acute stroke will be identified and offered the opportunity to participate in the study by research trained paramedics from the North East Ambulance Service NHS Trust. Patients who agree to participate in the study will receive either lisinopril (a common blood pressure lowering medication) or 'dummy' (placebo) treatments for seven days. The first dose of medication will be given by the paramedic in the ambulance. Subsequent tablets will be given in hospital. The effects of treatment will be monitored by measuring blood pressure, neurological outcome and adverse events.

All aspects of study feasibility including recruitment rates and compliance with data collection will be recorded. The study will run for one year and recruit 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 40 years old
* New unilateral arm weakness thought to be due to acute stroke within 3 hours of symptom onset
* Hypertension as defined by systolic BP >160mm Hg on two consecutive seated or lying readings taken 5 - 10 minutes apart
* Conscious (eyes open spontaneously ie "A" on Alert, Voice, Pain, Unresponsive (AVPU) scale)
* Patient being transported to a PIL-FAST trial site (i.e. Royal Victoria Infirmary, North Tyneside General Hospital and Wansbeck General Hospital)
* Verbal consent obtained from participant or next of kin

Exclusion criteria:

* Age < 40 years
* Females who are pregnant, lactating or at risk of pregnancy (i.e. who are not surgically sterile or at least 1 year post last menstrual period). Females < 56 years of age consented by a relative will be excluded as menstrual history may be unknown.
* Any presentation of suspected stroke without unilateral arm weakness
* Cannot establish that stroke onset time (i.e. when patient was last seen well without symptoms) was within the last 3 hours
* Systolic BP < 160mm Hg
* Reduced level of consciousness (below "A" on AVPU scale)
* Patient not being transported to PIL-FAST trial site
* Absence of participant or next of kin consent
* Known to be taking ACE-inhibitor or Angiotensin II Receptor Blocker medication already
* Known sensitivity to lisinopril or other ACE-inhibitor medication
* Pulse > 120 beats per minute
* Seizure activity in this illness episode (witnessed or history)
* Hypoglycaemia (blood glucose < 3.5 mmols/l)
* Cannot walk independently prior to stroke (walking stick / frame is allowed)
* Obvious understanding or memory problems when next of kin is absent
* Significant head trauma or brain surgery in the last 3 months
* Known renal failure
* Known liver failure (or currently jaundiced)
* Uncontrolled heart failure (breathlessness at rest)
* Receiving palliative care for known malignancy
* Currently enrolled in a clinical trial assessing a study drug

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of participants enrolled per month | 1 year
  The primary outcome measure is the number of participants enrolled in the study per month.

SECONDARY OUTCOMES:
Proportion fulfilling eligibility criteria | 1 year
  The proportion of suspected acute stroke patients admitted to research sites during the trial duration who fulfilled the study eligibility criteria
Proportion attended by research trained paramedic | 1 year
  The proportion of study eligible patients attended by a research trained paramedic
Proportion enrolled by research trained paramedic | 1 year
  The proportion of study eligible patients enrolled into the study by a researc trained paramedic
Proportion approached but not enrolled | 1 year
  The proportion of study eligible patients approached about the research study but not enrolled, and the reasons for non-enrolment, where possible.
Additional time spent on scene | 1 year
  The additional time spent on scene by research trained paramedics to enrol a participant into the study.
Paramedic compliance | 1 year
  Paramedic compliance with study data collection.
Hospital staff compliance | 1 year
  Hospital staff compliance with study medication administration and data collection.
Proportion completing study medication | 1 year
  The proportion of study participants with confirmed stroke who complete seven days of study medication.
Clinical outcome measures | 1 year
  Clinical outcome measures are blood pressure, neurological score, dependency score and renal function.
Adverse events | 1 year
  Adverse events in control and intervention groups during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Price, Principal Investigator — Northumbria Healthcare NHS Foundation Trust; Anand Dixit, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust; Ann Fox, Principal Investigator — North East Ambulance Service NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Wansbeck General Hospital, Ashington, Northumberland
  - Royal Victoria Infirmary, Queen Victoria Road, Newcastle upon Tyne, Tyne and Wear
  - North East Ambulance Service NHS Trust, Newcastle upon Tyne, Tyne and Wear
  - North Tyneside General Hospital, North Shields, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No
No IPD were shared, nor will be, from this trial.

REFERENCES:
- [Derived] Shaw L, Price C, McLure S, Howel D, McColl E, Younger P, Ford GA. Paramedic Initiated Lisinopril For Acute Stroke Treatment (PIL-FAST): results from the pilot randomised controlled trial. Emerg Med J. 2014 Dec;31(12):994-9. doi: 10.1136/emermed-2013-202536. Epub 2013 Sep 27. PMID 24078198
- [Derived] Shaw L, Price C, McLure S, Howel D, McColl E, Ford GA. Paramedic Initiated Lisinopril For Acute Stroke Treatment (PIL-FAST): study protocol for a pilot randomised controlled trial. Trials. 2011 Jun 15;12:152. doi: 10.1186/1745-6215-12-152. PMID 21676221